CLINICAL TRIAL: NCT06804070
Title: Clinical and Instrumental Efficacy Evaluation on Eczema of One Cosmetic Product
Brief Title: The Effects of a Botanical Moisturizer and an Unscented Soap on Eczema and Itch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Codex Labs Corporation (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #STUU524AA0147-1
Record Dates: First submitted 2025-01-12; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis (Eczema)
Keywords: eczema; skin care; botanical; dry skin; itch
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant (Experimental): The participant is provided with and instructed to use a botanical moisturizer on the body for the duration of the study. The participant is also provided with and instructed to use an unscented soap, in replacement of the participant's usual cleansing product for the duration of the study.
  Interventions: Other: Botanical Moisturizer + Unscented Soap

INTERVENTIONS:
Other: Botanical Moisturizer + Unscented Soap — The intervention includes the use of 2 products:
  1. A botanical moisturizer
  2. An unscented bar of soap

SUMMARY:
The purpose of this study is to examine the effects of a botanical moisturizer and an unscented soap on eczema severity, itch, mood, and various skin measures (such as skin hydration) in those with mild to moderate eczema.

ELIGIBILITY:
Inclusion Criteria:

* Sex: female and male;
* Age : 18 years old and above;
* Phototype: I to IV;
* Type: Caucasian;
* Subjects with active eczema condition the body (showing flakiness, irritation, itch and intense dryness);
* Subjects with a SCORAD of 25 - 50;
* Subjects with dry skin on the study areas;
* Subject barely wearing makeup;
* Subjects must not take antibiotics and / or apply any antifungal treatments (body/scalp) for 1 month before study start and during the entire study duration;
* No change in hygiene, cosmetics, and make-up habits - except for the product(s) under study - during the entire study duration;
* Subjects agreeing not to change lifestyle habits during the study duration.
* Healthy subject;
* Subject having given her free informed, written consent;
* Subject willing to adhere to the protocol and study procedures;
* Subject with Polish citizenship.

Exclusion Criteria:

* For women with childbearing potential: pregnant or nursing woman or woman planning to get pregnant during the study;
* Cutaneous pathology on the study zone (other than eczema);
* Use of topical or systemic treatment during the previous weeks liable to interfere with the assessment of the study product (the subjects are allowed to use their topical corticosteroids during the study if needed; the information about the treatment and the number of applications must be noted in the daily log);
* Subject having undergone a surgery under general anesthesia within the previous month;
* Excessive exposure to sunlight or UV-rays within the previous month;
* Subject enrolled in another clinical trial during the study period (concerns the studied zones).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Objective and Subjective Scoring of Eczema Severity | 8 weeks
  Change in eczema severity was assessed using SCORAD (SCOring of Atopic Dermatitis).
  A. First, the spread of eczema on different body areas is assessed by the investigator and calculated as a percent, where the maximum is 100%.
  B. Second, the intensity of skin redness, swelling, oozing, scratch marks, skin thickening and dryness is scored by the investigator from 0 to 3, where 0 is none, 1 is mild, 2 is moderate, and 3 is severe.
  C. Finally, for the subjective score, participants are asked to report the intensity of symptoms (itch and sleeplessness) from 0 to 10, where 0 is no itch or no sleeplessness, and 10 is the worst imaginable itch or insomnia sleeplessness.
  The total score of the objective SCORAD is obtained with the following formula:
  SCORAD = A/5 + 7 B/2 + C
Localized Eczema Severity | 4 weeks
  Change in localized eczema severity is assessed with the Eczema Area and Severity Index (EASI).
  Skin redness, elevation, scratching, and thickening are assessed by the investigator on a scale of 0 to 3, where 0 is none, 1 is mild, 2 is moderate, 3 is severe. The localized EASI is the sum of these scores.
Localized Eczema Severity | 8 weeks
  Change in localized eczema severity is assessed with the Eczema Area and Severity Index (EASI).
  Skin redness, elevation, scratching, and thickening are assessed by the investigator on a scale of 0 to 3, where 0 is none, 1 is mild, 2 is moderate, 3 is severe. The localized EASI is the sum of these scores.

SECONDARY OUTCOMES:
Skin Hydration | 4 weeks
  Change in skin hydration is assessed with a Corneometer.
Skin Hydration | 8 weeks
  Change in skin hydration is assessed with a Corneometer.
Transepidermal Water Loss | 4 weeks
  Change in transepidermal water loss is assessed with a Tewameter TM 300
Transepidermal Water Loss | 8 weeks
  Change in transepidermal water loss is assessed with a Tewameter TM 300
Desquamation Index | 4 weeks
  Change in desquamation is assessed with D-Squam®.
Desquamation Index | 8 weeks
  Change in desquamation is assessed with D-Squam®.
Positive and Negative Affect | 4 weeks
  Change in mood is assessed with the PANAS-SF (Positive and Negative Affect Schedule- Short Form).
  Participants are asked to evaluate the degree to which they experienced components of positive and negative affect : Interested, Distressed, Excited, Upset, Strong, Guilty, Scared, Hostile, Enthusiastic, Proud, Irritable, Alert, Ashamed, Inspired, Nervous, Determined, Attentive, Jittery, Active, and Afraid. A 5-point scale was used where 1 is very slightly or not at all, 2 is a little, 3 is moderately, 4 is quite a bit, and 5 is extremely.
Positive and Negative Affect | 8 weeks
  Change in mood is assessed with the PANAS-SF (Positive and Negative Affect Schedule- Short Form).
  Participants are asked to evaluate the degree to which they experienced components of positive and negative affect : Interested, Distressed, Excited, Upset, Strong, Guilty, Scared, Hostile, Enthusiastic, Proud, Irritable, Alert, Ashamed, Inspired, Nervous, Determined, Attentive, Jittery, Active, and Afraid. A 5-point scale was used where 1 is very slightly or not at all, 2 is a little, 3 is moderately, 4 is quite a bit, and 5 is extremely.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermscan Poland, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No
Data will need to be protected for patentability reasons while IP is being filed. Once IP considerations are finalized, data can be shared.